CLINICAL TRIAL: NCT04539496
Title: A Multicenter, Open-label Phase I/II Study of XZP-3287 in Metastasis Solid Tumors in China
Brief Title: A Phase I/II Study of XZP-3287 in Metastasis Solid Tumors
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Sihuan Pharmaceutical Holdings Group Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: XZP-3287-1001
Record Dates: First submitted 2020-08-26; First posted 2020-09-07 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Metastasis Solid Tumors; Advanced Breast Cancer

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Dose Escalation and Expansion Study (Experimental): To determine the MTD and RP2D of XZP-3287
  Interventions: Drug: XZP-3287
- Combination Therapy Study (Experimental): To determine the RP2D of XZP-3287 combined with endocrine therapy
  Interventions: Drug: XZP-3287;Letrozole;Anastrozole;Fulvestrant
- A Phase 2 Study of Single-Agent XZP-3287 in Patients After Failure of Multi-Line Therapy (Experimental): To determine the efficacy and safety profiles of XZP-3287 as a single- agent in hormone receptor (HR) positive, human epidermal growth factor receptor 2 (HER2) negative advanced breast cancer
  Interventions: Drug: XZP-3287

INTERVENTIONS:
Drug: XZP-3287 — * 20-560 mg QD, oral
  * 240-480 mg BID, oral
  Arms: Dose Escalation and Expansion Study
Drug: XZP-3287;Letrozole;Anastrozole;Fulvestrant — XZP-3287: 360 mg BID, oral; Letrozole: 2.5 mg QD, oral; Anastrozole: 1 mg QD, oral; Fulvestrant: 500 mg intramuscular injection on C1D1, C1D15, the first day of each subsequent cycle (28 days a cycle)
  Arms: Combination Therapy Study
Drug: XZP-3287 — 480 mg BID, oral
  Arms: A Phase 2 Study of Single-Agent XZP-3287 in Patients After Failure of Multi-Line Therapy

SUMMARY:
This study includes single agent/combination dose exploration study and the phase II study. The primary purpose of the dose exploration study is to determine the maximum tolerated dose(MTD)/recommended phase II dose(RP2D) of XZP-3287 and assess its safety and preliminary efficacy in solid tumor patients. The phase II study aims to explore the efficacy and safety profiles of XZP-3287 as a single- agent in hormone receptor(HR) positive, human epidermal growth factor receptor 2(HER2) negative advanced breast cancer.

ELIGIBILITY:
Inclusion Criteria:

* Single agent and combination dose exploration study：Patient is an adult male/female 18~70 years old; the phase II study：Patient is an adult male/female ≥ 18 years old;
* Single agent dose escalation study ：Patients with a histologically or cytologically confirmed diagnosis of a solid tumor for which Standard treatment failure or no further effective standard treatment is available.

Combination dose exploration study：Patients with locally advanced or metastatic breast cancer with hormone receptor positive (HR+) and her2-negative (HER2-) were not eligible for surgical resection or radiotherapy for the purpose of cure, and had no clinical indications for chemotherapy, and received endocrine therapy ≤1 line.

The phase II study: Locally advanced or metastatic breast cancer diagnosed histologically or cytologically not suitable for surgery or radical radiotherapy; HR+ and HER2- ; have locally advanced disease not amenable to curative treatment by surgery or metastatic disease; progress after previous endocrine therapy; at least 1 chemotherapy regimen in the previous adjuvant or metastasis contains paclitaxel; there should be at least 2 prior chemotherapy regimens;

* At least one measurable lesion (based on RECIST v1.1);
* Patient has an Eastern Cooperative Oncology Group (ECOG) performance status 0 or 1;
* Have recovered from the acute effects of therapy (until the toxicity resolves to either baseline or Grade 1) except for residual alopecia;
* Adequate organ and marrow function;
* The life expectancy of the patient was determined by the investigator to be ≥12 weeks;
* Fertile male or female patients must agree to use an effective contraceptive method during the study period and for three months after the last study medication;
* Patient has signed informed consent before any trial related activities.

Exclusion Criteria:

* Single agent and combination dose exploration study：Patients with known uncontrolled or symptomatic CNS metastases; The phase II study：Have central nervous system (CNS) metastasis, or Have visceral crisis, or Inflammatory breast cancer.
* Have received an autologous or allogeneic stem-cell transplant.
* Patient has impairment of gastrointestinal (GI) function or GI disease.
* Single agent and combination dose exploration study：Any other malignancy was diagnosed within 3 years prior to enrollment, except for basal cell carcinoma, squamous cell carcinoma, or carcinoma in situ of the cervix, which is adequately treated and the disease is stable.

The phase II study：Have a history of any other cancer (except nonmelanoma skin cancer or carcinoma in-situ of the cervix), unless in complete remission with no therapy for a minimum of 3 years.

* Subject has impaired cardiac function or heart disease of clinical significance.
* Cerebrovascular accidents within 6 months before enrollment, including a history of transient ischemic attack or stroke.
* Major surgery or surgical treatment due to any cause occurred within 4 weeks prior to enrollment.
* Presence of any serious and/or uncontrolled disease in the opinion of the investigator that may interfere with the study assessment.
* Uncontrollable pleural effusion, peritoneal effusion, pericardial effusion in the 4 weeks before the first administration (except for a small amount of effusion detected by imaging examination).
* A prior history of definite neurological or psychiatric disorders, including epilepsy or dementia.
* Chronic active HBV, HCV or HIV diseases.
* Patient who received any CDK4/6 inhibitor or patients who plan surgery, or the investigator determines that surgery or radical radiation therapy is required.
* Participation in a prior treatment of chemotherapy, radiotherapy, endocrinotherapy, targeted therapy, immunotherapy and any investigational study within 14 days prior to enrollment.
* Bone marrow suppression therapy, such as GCS-F, EPO, or blood transfusion, was administered within 14 days prior to enrollment.
* Patient with a known hypersensitivity to any of the excipients in this study.
* Pregnant or breastfeeding.
* The researchers considered that there were some cases that were not suitable for inclusion.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 402 (Actual)
Dates: Start 2018-05-22 (Actual); Primary Completion 2023-07-31 (Actual); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Single agent and combination dose exploration study：AE evaluation | Up to 30 days after the end of treatment
  AEs as characterized by frequency and severity (as graded by National Cancer Institute Common Terminology Criteria for Adverse Events [NCI CTCAE] version 4.03 for single agent dose exploration study and CTCAE 5.0 for combination exploration study)
The phase II study：Objective response rate (ORR) assessed by Independent Review Committee (IRC) | From baseline to the date of first documentation of progression or death , whichever came first, assessed approximately up to 2 years after the last entered participant
  ORR is the percentage of participants with a best overall response (BOR) of complete response (CR) or partial response (PR) as defined by RECIST v1.1.

SECONDARY OUTCOMES:
Progression free survival (PFS) | From baseline to the date of first documentation of progression or death, whichever came first, assessed approximately up to 2 years after the last entered participant
  PFS is defined as the time from the date of the first treatment until first observation of objective progressive disease or death, whichever comes first.
Overall survival (OS) | From baseline to the death from any cause, assessed approximately up to 2 years after the last entered participant
  OS is defined from the date of the first treatment to the date of death from any cause.
Duration of response (DoR) | From baseline to the date of first documentation of progression or death, whichever came first, assessed approximately up to 2 years after the last entered participant
  DoR is defined from the date of CR or PR to date of disease progression or death due to any cause.
Disease control rate (DCR) | From baseline to the date of first documentation of progression or death, whichever came first, assessed approximately up to 2 years after the last entered participant
  DCR is the percentage of participants with a best overall response of CR, PR or stable disease (SD) as defined by RECIST v1.1.
Clinical benefit rate (CBR) | From baseline to the date of first documentation of progression or death, whichever came first, assessed approximately up to 2 years after the last entered participant
  Percentage of participants with best overall response of CR, PR, or SD with duration of SD for at least 6 Months.
Pharmacokinetics (PK) | From baseline up to month 3
  Mean steady state exposure of XZP-3287 and its metabolites.
Investigator-assessed ORR | From baseline to the date of first documentation of progression or death, whichever came first, assessed approximately up to 2 years after the last entered participant
  ORR is the percentage of participants with a best overall response (BOR) of complete response (CR) or partial response (PR) as defined by RECIST v1.1.
The phase II study：AE evaluation | Up to 30 days after the end of treatment
  AEs as characterized by frequency and severity (as graded by CTCAE 5.0 )

CONTACTS AND LOCATIONS:
Locations (1):
- Cancer Hospital Chinese Academy of Medical Sciences, Beijing, Beijing Municipality, China

REFERENCES:
- [Derived] Wang J, Sun T, Tong Z, Hu X, Li W, Yan M, Liu Y, Ouyang Q, Liu X, Fang J, Li H, Li H, Chen W, Gong C, Teng Y, Xu L, Duan X, Liu M, Meng Y, Liu F, Wang L, Xu B. Safety and tolerability of bireociclib for the treatment of advanced solid tumors as monotherapy and in combination with endocrine therapy: a multicenter, open-label, phase 1 clinical trial. BMC Med. 2025 Oct 8;23(1):546. doi: 10.1186/s12916-025-04364-9. PMID 41063198
- [Derived] Wang J, Zhang Q, Sun T, Li H, Cheng Y, Tong Z, Li H, Li W, Wang J, Teng Y, Wu X, Cheng J, Chen Z, Zhu Z, Wang L, Liu M, Duan X, Xu L, Xu B. An open-label, single-arm, multicenter, phase II trial of bireociclib as monotherapy for heavily pretreated HR-positive, HER2-negative advanced breast cancer patients: BRIGHT-1 trial. Cancer Commun (Lond). 2025 Jun;45(6):640-653. doi: 10.1002/cac2.70009. Epub 2025 Feb 27. PMID 40013319